CLINICAL TRIAL: NCT02662569
Title: A Double-blind, Randomized, Placebo-controlled, Multicenter Study to Evaluate Safety and Efficacy of Evolocumab (AMG 145) in Combination With Statin Therapy in Diabetic Subjects With Hyperlipidemia or Mixed Dyslipidemia (BERSON)
Brief Title: Safety and Efficacy of Evolocumab in Combination With Statin Therapy in Adults With Diabetes and Hyperlipidemia or Mixed Dyslipidemia
Acronym: BERSON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20120119; 2013-000723-14 (EudraCT Number)
Record Dates: First submitted 2016-01-20; First posted 2016-01-25 (Estimated); Results first posted 2019-01-11 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Diabetes, Hyperlipidemia, Mixed Dyslipidemia
MeSH Terms: conditions — Diabetes Mellitus; Hyperlipidemias | interventions — evolocumab; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Atorvastatin (Q2W) (Active Comparator): Participants received placebo subcutaneous injection once every 2 weeks (Q2W) and 20 mg atorvastatin orally once a day for up to 12 weeks.
  Interventions: Drug: Atorvastatin; Other: Placebo
- Atorvastatin (QM) (Active Comparator): Participants received placebo subcutaneous injection once a month (QM) and 20 mg atorvastatin orally once a day for up to 12 weeks.
  Interventions: Drug: Atorvastatin; Other: Placebo
- Evolocumab Q2W + Atorvastatin (Experimental): Participants received 140 mg evolocumab by subcutaneous injection once every 2 weeks and 20 mg atorvastatin orally once a day for up to 12 weeks.
  Interventions: Biological: Evolocumab; Drug: Atorvastatin
- Evolocumab QM + Atorvastatin (Experimental): Participants received 420 mg evolocumab by subcutaneous injection once a month and 20 mg atorvastatin orally once a day for up to 12 weeks.
  Interventions: Biological: Evolocumab; Drug: Atorvastatin

INTERVENTIONS:
Biological: Evolocumab — Administered by subcutaneous injection
  Other Names: AMG 145; Repatha
  Arms: Evolocumab Q2W + Atorvastatin; Evolocumab QM + Atorvastatin
Drug: Atorvastatin — Administered orally once a day
  Other Names: Lipitor
Other: Placebo — Placebo to evolocumab administered by subcutaneous injection
  Arms: Atorvastatin (Q2W); Atorvastatin (QM)

SUMMARY:
The primary objective of this study was to evaluate the effect of 12 weeks of subcutaneous evolocumab (AMG 145) in combination with statin therapy (atorvastatin) on percent change from baseline in low-density lipoprotein cholesterol (LDL-C) in diabetic adults with hyperlipidemia or mixed dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with type 2 diabetes (receiving pharmacologic treatment for at least 6 months or longer) with stable diabetes therapy
* Lipid-lowering therapy must be unchanged for at least 4 weeks or more
* Subjects receiving statin therapy at screening must have a fasting LDL-C of greater than or equal to 100 mg/dL
* Subjects not receiving statin therapy at screening must have a fasting LDL-C of greater than or equal to 130 mg/dL

Exclusion criteria:

* New York Heart Association (NYHA) class III or IV heart failure
* Uncontrolled cardiac arrhythmia
* Uncontrolled hypertension
* Type 1 diabetes or poorly controlled type 2 diabetes
* Uncontrolled hypothyroidism or hyperthyroidism.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 986 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2017-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (79):
- United States (11):
  - Research Site, Miami, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Indianapolis, Indiana
  - Research Site, Iowa City, Iowa
  - Research Site, Overland Park, Kansas
  - Research Site, Monroe, Louisiana
  - Research Site, St Louis, Missouri
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Dallas, Texas
  - Research Site, San Antonio, Texas
- Argentina (5):
  - Research Site, CABA, Buenos Aires
  - Research Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Research Site, Mar del Plata, Buenos Aires
  - Research Site, Buenos Aires
  - Research Site, Córdoba
- Brazil (4):
  - Research Site, Brasília, Federal District
  - Research Site, Goiânia, Goiás
  - Research Site, São Paulo, São Paulo
  - Research Site, Rio de Janeiro
- Canada (8):
  - Research Site, Winnipeg, Manitoba
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Woodstock, Ontario
  - Research Site, Laval, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Saint-Jean-sur-Richelieu, Quebec
  - Research Site, Sherbrooke, Quebec
- China (31):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Chongqing, Chongqing Municipality
  - Research Site, Guangzhou, Guangdong
  - Research Site, Nanning, Guangxi
  - Research Site, Guiyang, Guizhou
  - Research Site, Shijiazhuang, Hebei
  - Research Site, Wuhan, Hubei
  - Research Site, Changsha, Hunan
  - Research Site, Hengyang, Hunan
  - Research Site, Zhuzhou, Hunan
  - Research Site, Baotou, Inner Mongolia
  - Research Site, Nanjing, Jiangsu
  - Research Site, Suzhou, Jiangsu
  - Research Site, Wuxi, Jiangsu
  - Research Site, Xuzhou, Jiangsu
  - Research Site, Zhenjiang, Jiangsu
  - Research Site, Nanchang, Jiangxi
  - Research Site, Changchun, Jilin
  - Research Site, Siping, Jilin
  - Research Site, Shenyang, Liaoning
  - Research Site, Xi'an, Shaanxi
  - Research Site, Jinan, Shandong
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Chengdu, Sichuan
  - Research Site, Tianjin, Tianjin Municipality
  - Research Site, Ürümqi, Xinjiang
  - Research Site, Hangzhou, Zhejiang
  - Research Site, Linhai, Zhejiang
  - Research Site, Wenzhou, Zhejiang
  - Research Site, Beijing
  - Research Site, Shanghai
- Colombia (3):
  - Research Site, Medellín, Antioquia
  - Research Site, Barranquilla, Atlántico
  - Research Site, Pasto, Departamento de Nariño
- France (3):
  - Research Site, Dijon
  - Research Site, Nantes
  - Research Site, Toulouse
- Russia (5):
  - Research Site, Kemerovo
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Tomsk
- South Korea (5):
  - Research Site, Bucheon-si, Wonmi-gu
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Turkey (Türkiye) (4):
  - Research Site, Antalya
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Kocaeli

REFERENCES:
- [Derived] Blom DJ, Chen J, Yuan Z, Borges JLC, Monsalvo ML, Wang N, Hamer AW, Ge J. Effects of evolocumab therapy and low LDL-C levels on vitamin E and steroid hormones in Chinese and global patients with type 2 diabetes. Endocrinol Diabetes Metab. 2020 Mar 6;3(2):e00123. doi: 10.1002/edm2.123. eCollection 2020 Apr. PMID 32318641
- [Derived] Chen Y, Yuan Z, Lu J, Eliaschewitz FG, Lorenzatti AJ, Monsalvo ML, Wang N, Hamer AW, Ge J. Randomized study of evolocumab in patients with type 2 diabetes and dyslipidaemia on background statin: Pre-specified analysis of the Chinese population from the BERSON clinical trial. Diabetes Obes Metab. 2019 Jun;21(6):1464-1473. doi: 10.1111/dom.13700. Epub 2019 Apr 14. PMID 30851062
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 102 study centers and randomized at 98 centers in Argentina, Brazil, Canada, China, Colombia, France, Republic of Korea, Russian Federation, Turkey, and the United States from 14 April 2016 to 28 July 2017.
Pre-assignment Details: Participants who met eligibility criteria and completed at least 4 weeks of lipid stabilization on atorvastatin 20 mg daily were randomized in a 1:1:2:2 ratio to receive placebo every 2 weeks (Q2W), placebo once a month (QM), evolocumab Q2W, or evolocumab QM. Randomization was stratified by entry statin therapy and geographic region.
Groups:
- Placebo Q2W: Participants received placebo subcutaneous injection once every 2 weeks (Q2W) and 20 mg atorvastatin orally once a day for up to 12 weeks.
- Placebo QM: Participants received placebo subcutaneous injection once a month (QM) and 20 mg atorvastatin orally once a day for up to 12 weeks.
- Evolocumab Q2W: Participants received 140 mg evolocumab by subcutaneous injection once every 2 weeks and 20 mg atorvastatin orally once a day for up to 12 weeks.
- Evolocumab QM: Participants received 420 mg evolocumab by subcutaneous injection once a month and 20 mg atorvastatin orally once a day for up to 12 weeks.
Period: Overall Study
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Started | 166 | 161 | 327 | 332
Received Study Drug (Study drug defined as subcutaneous evolocumab or placebo to evolocumab) | 164 | 160 | 325 | 332
Completed | 159 | 160 | 321 | 328
Not Completed | 7 | 1 | 6 | 4
Not completed — Withdrawal by Subject | 6 | 1 | 6 | 4
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM | Total
Number analyzed (Participants) | 166 | 161 | 327 | 332 | 986
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (8.8) | 61.0 (8.8) | 61.0 (8.5) | 61.6 (8.4) | 61.3 (8.6)
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 years | 105 | 101 | 206 | 208 | 620
  65 - 80 years | 61 | 60 | 121 | 124 | 366
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 94 | 178 | 190 | 564
  Male | 64 | 67 | 149 | 142 | 422
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 34 | 65 | 67 | 195
  Not Hispanic or Latino | 137 | 127 | 262 | 265 | 791
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 0 | 2
  Asian | 82 | 80 | 164 | 166 | 492
  Black or African American | 7 | 6 | 11 | 18 | 42
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  White | 72 | 68 | 140 | 140 | 420
  Multiple | 5 | 6 | 11 | 8 | 30
Stratification Factor: Statin Therapy at Study Entry [Count of Participants; unit: Participants] — Intensive: at least one of the following recorded for the last 4 weeks prior to screening: atorvastatin ≥ 40 mg once daily (QD); rosuvastatin ≥ 20 mg QD; simvastatin ≥ 80 mg QD; any statin (atorvastatin, fluvastatin, lovastatin, pitavastatin, pravastatin, rosuvastatin, and simvastatin) QD plus ezetimibe.
  Non-intensive: Participant was taking any dose of a statin at least weekly for the last 4 weeks prior to screening and is not included in the intensive statin usage.
  No statin: Participant was not included in the intensive statin usage or non-intensive statin usage.
  Participants
    Intensive statin usage | 16 | 15 | 31 | 32 | 94
    Non-intensive statin usage | 83 | 80 | 167 | 166 | 496
    No statin | 67 | 66 | 129 | 134 | 396
Stratification Factor: Geographic Region [Count of Participants; unit: Participants]
  China | 76 | 75 | 150 | 152 | 453
  South Korea | 6 | 5 | 14 | 13 | 38
  Other countries | 84 | 81 | 163 | 167 | 495
Low-density Lipoprotein Cholesterol (LDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] — Population: Full analysis set, defined as all randomized participants who received at least 1 dose of study drug (subcutaneous evolocumab or placebo to evolocumab).
  mg/dL
    number analyzed (Participants) | 164 | 160 | 325 | 332 | 981
    (all) | 92.2 (32.0) | 91.0 (30.7) | 92.4 (33.8) | 93.5 (33.6) | 92.5 (32.9)
Non-high-density Lipoprotein Cholesterol (non-HDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] — Population: Full analysis set
  mg/dL
    number analyzed (Participants) | 164 | 160 | 325 | 332 | 981
    (all) | 119.2 (38.2) | 119.4 (36.0) | 121.3 (38.1) | 121.2 (37.0) | 120.6 (37.4)
Apolipoprotein B100 Concentration [Mean (Standard Deviation); unit: mg/dL] — Apolipoprotein B100 is the primary apolipoprotein of low-density lipoprotein cholesterol particles, and plays a role in moving cholesterol around the body. Population: Full analysis set with available data
  mg/dL
    number analyzed (Participants) | 162 | 158 | 325 | 332 | 977
    (all) | 82.1 (23.1) | 83.4 (22.3) | 84.8 (23.0) | 84.4 (21.8) | 84.0 (22.5)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] — Population: Full analysis set
  mg/dL
    number analyzed (Participants) | 164 | 160 | 325 | 332 | 981
    (all) | 166.5 (38.6) | 169.3 (37.5) | 167.8 (38.9) | 168.9 (38.9) | 168.2 (38.6)
Total Cholesterol/High-density Lipoprotein Cholesterol(HDL-C) Ratio [Mean (Standard Deviation); unit: ratio] — Population: Full analysis set
  ratio
    number analyzed (Participants) | 164 | 160 | 325 | 332 | 981
    (all) | 3.717 (1.337) | 3.598 (1.071) | 3.804 (1.273) | 3.725 (1.201) | 3.729 (1.229)
Apolipoprotein B100/Apolipoprotein A1 Ratio [Mean (Standard Deviation); unit: ratio] — Population: Full analysis set with available data
  ratio
    number analyzed (Participants) | 162 | 158 | 325 | 332 | 977
    (all) | 0.573 (0.192) | 0.563 (0.161) | 0.601 (0.200) | 0.586 (0.185) | 0.585 (0.188)
Lipoprotein (a) [Mean (Standard Deviation); unit: nmol/L] — Population: Full analysis set
  nmol/L
    number analyzed (Participants) | 164 | 160 | 325 | 332 | 981
    (all) | 67.0 (90.9) | 71.8 (96.5) | 65.6 (92.5) | 73.2 (95.9) | 69.4 (94.0)
Triglycerides Concentration [Mean (Standard Deviation); unit: mg/dL] — Population: Full analysis set
  mg/dL
    number analyzed (Participants) | 164 | 160 | 325 | 332 | 981
    (all) | 137.3 (77.3) | 150.6 (154.6) | 145.9 (67.5) | 139.7 (64.9) | 143.1 (88.4)
High-density Lipoprotein Cholesterol (HDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] — Population: Full analysis set
  mg/dL
    number analyzed (Participants) | 164 | 160 | 325 | 332 | 981
    (all) | 47.3 (11.9) | 49.9 (15.2) | 46.5 (11.5) | 47.6 (12.3) | 47.6 (12.6)
Very Low-density Lipoprotein Cholesterol (VLDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] — Population: Full analysis set
  mg/dL
    number analyzed (Participants) | 164 | 160 | 325 | 332 | 981
    (all) | 27.3 (14.9) | 28.4 (16.2) | 28.7 (12.6) | 27.8 (12.7) | 28.1 (13.7)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in LDL-C at the Mean of Weeks 10 and 12
Time Frame: Baseline and weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 164 | 160 | 325 | 332
percent change | 4.94 (3.48) | 0.99 (3.31) | -65.35 (3.09) | -69.05 (2.96)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; The model includes treatment group, entry statin therapy and geographic region, scheduled visit, and the interaction of treatment with scheduled visit; LS Mean Treatment Difference = -70.29, 95% CI 2-sided [-75.43 to -65.16], Standard Error of Mean 2.61 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -70.04, 95% CI 2-sided [-74.67 to -65.41], Standard Error of Mean 2.35 — Treatment difference = Evolocumab QM - Placebo QM

2. Primary Outcome: Percent Change From Baseline in LDL-C at Week 12
Time Frame: Baseline and week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 164 | 160 | 325 | 332
percent change | 7.10 (3.66) | 2.63 (3.41) | -64.66 (3.20) | -62.30 (3.02)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -71.77, 95% CI 2-sided [-77.61 to -65.93], Standard Error of Mean 2.97 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -64.93, 95% CI 2-sided [-69.97 to -59.89], Standard Error of Mean 2.56 — Treatment difference = Evolocumab QM - Placebo QM

3. Secondary Outcome: Change From Baseline in LDL-C at the Mean of Weeks 10 and 12
Time Frame: Baseline and weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 164 | 160 | 325 | 332
mg/dL | -2.1 (4.1) | -8.8 (4.0) | -64.6 (3.6) | -71.9 (3.6)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -62.5, 95% CI 2-sided [-68.2 to -56.9], Standard Error of Mean 2.9 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -63.1, 95% CI 2-sided [-68.4 to -57.8], Standard Error of Mean 2.7 — Treatment difference = Evolocumab QM - Placebo QM

4. Secondary Outcome: Change From Baseline in LDL-C at Week 12
Time Frame: Baseline and week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 164 | 160 | 325 | 332
mg/dL | -0.3 (4.2) | -7.3 (4.1) | -63.9 (3.7) | -66.1 (3.7)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -63.6, 95% CI 2-sided [-69.7 to -57.6], Standard Error of Mean 3.1 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -58.8, 95% CI 2-sided [-64.3 to -53.3], Standard Error of Mean 2.8 — Treatment difference = Evolocumab QM - Placebo QM

5. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at the Mean of Weeks 10 and 12
Time Frame: Baseline and weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 164 | 160 | 325 | 332
percent change | 4.33 (3.05) | 0.33 (2.95) | -56.57 (2.70) | -59.08 (2.63)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -60.90, 95% CI 2-sided [-65.51 to -56.29], Standard Error of Mean 2.35 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -59.40, 95% CI 2-sided [-63.52 to -55.29], Standard Error of Mean 2.09 — Treatment difference = Evolocumab QM - Placebo QM

6. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 12
Time Frame: Baseline and week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 164 | 160 | 325 | 332
percent change | 5.87 (3.20) | 1.30 (3.03) | -55.76 (2.79) | -52.92 (2.69)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -61.64, 95% CI 2-sided [-66.82 to -56.45], Standard Error of Mean 2.64 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -54.22, 95% CI 2-sided [-58.70 to -49.74], Standard Error of Mean 2.28 — Treatment difference = Evolocumab QM - Placebo QM

7. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B100 at the Mean of Weeks 10 and 12
Time Frame: Baseline and weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 164 | 160 | 325 | 332
percent change | 1.97 (3.31) | -1.52 (2.99) | -54.96 (3.07) | -56.37 (2.72)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -56.93, 95% CI 2-sided [-60.93 to -52.93], Standard Error of Mean 2.03 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -54.85, 95% CI 2-sided [-58.52 to -51.18], Standard Error of Mean 1.87 — Treatment difference = Evolocumab QM - Placebo QM

8. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B100 at Week 12
Time Frame: Baseline and week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 164 | 160 | 325 | 332
percent change | 3.17 (3.42) | -0.26 (3.03) | -53.90 (3.14) | -49.68 (2.75)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -57.06, 95% CI 2-sided [-61.59 to -52.54], Standard Error of Mean 2.30 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -49.42, 95% CI 2-sided [-53.31 to -45.53], Standard Error of Mean 1.98 — Treatment difference = Evolocumab QM - Placebo QM

9. Secondary Outcome: Percent Change From Baseline in Total Cholesterol at the Mean of Weeks 10 and 12
Time Frame: Baseline and weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 164 | 160 | 325 | 332
percent change | 2.89 (2.30) | -0.25 (2.18) | -38.64 (2.04) | -39.74 (1.95)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -41.53, 95% CI 2-sided [-44.95 to -38.10], Standard Error of Mean 1.74 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -39.50, 95% CI 2-sided [-42.47 to -36.53], Standard Error of Mean 1.51 — Treatment difference = Evolocumab QM - Placebo QM

10. Secondary Outcome: Percent Change From Baseline in Total Cholesterol at Week 12
Time Frame: Baseline and week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 164 | 160 | 325 | 332
percent change | 4.40 (2.40) | 0.67 (2.24) | -37.82 (2.10) | -35.22 (1.99)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -42.22, 95% CI 2-sided [-46.02 to -38.42], Standard Error of Mean 1.93 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -35.89, 95% CI 2-sided [-39.12 to -32.67], Standard Error of Mean 1.64 — Treatment difference = Evolocumab QM - Placebo QM

11. Secondary Outcome: Percent Change From Baseline in Total Cholesterol/HDL-C Ratio at the Mean of Weeks 10 and 12
Time Frame: Baseline and weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 164 | 160 | 325 | 332
percent change | 3.03 (2.38) | -2.03 (2.41) | -41.06 (2.11) | -45.70 (2.17)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -44.09, 95% CI 2-sided [-47.64 to -40.54], Standard Error of Mean 1.81 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -43.67, 95% CI 2-sided [-46.90 to -40.44], Standard Error of Mean 1.64 — Treatment difference = Evolocumab QM - Placebo QM

12. Secondary Outcome: Percent Change From Baseline in Total Cholesterol/HDL-C Ratio at Week 12
Time Frame: Baseline and week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 164 | 160 | 325 | 332
percent change | 3.22 (2.49) | -1.22 (2.47) | -40.72 (2.18) | -41.78 (2.21)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -43.94, 95% CI 2-sided [-47.90 to -39.97], Standard Error of Mean 2.02 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -40.56, 95% CI 2-sided [-44.08 to -37.04], Standard Error of Mean 1.79 — Treatment difference = Evolocumab QM - Placebo QM

13. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B100/Apolipoprotein A1 Ratio at the Mean of Weeks 10 and 12
Time Frame: Baseline and weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 164 | 160 | 325 | 332
percent change | 2.60 (3.30) | -1.02 (3.09) | -55.60 (3.07) | -57.75 (2.82)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -58.20, 95% CI 2-sided [-62.15 to -54.25], Standard Error of Mean 2.01 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -56.73, 95% CI 2-sided [-60.53 to -52.93], Standard Error of Mean 1.93 — Treatment difference = Evolocumab QM - Placebo QM

14. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B100/Apolipoprotein A1 Ratio at Week 12
Time Frame: Baseline and week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 164 | 160 | 325 | 332
percent change | 3.23 (3.39) | -0.10 (3.16) | -54.98 (3.12) | -51.80 (2.86)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -58.21, 95% CI 2-sided [-62.59 to -53.84], Standard Error of Mean 2.23 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -51.70, 95% CI 2-sided [-55.81 to -47.59], Standard Error of Mean 2.09 — Treatment difference = Evolocumab QM - Placebo QM

15. Secondary Outcome: Percentage of Participants With Mean LDL-C at Weeks 10 and 12 of Less Than 70 mg/dL (1.8 mmol/L)
Time Frame: Weeks 10 and 12
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 164 | 160 | 325 | 332
percentage of participants | 21.7 [15.9 to 28.7] | 19.4 [13.9 to 26.3] | 90.1 [86.2 to 92.9] | 91.3 [87.6 to 93.9]
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Cochran-Mantel Haenszel test stratified by entry statin therapy and geographic region; Treatment Difference = 68.4, 95% CI 2-sided [60.4 to 74.8] — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Cochran-Mantel Haenszel test stratified by entry statin therapy and geographic region; Treatment Difference = 71.9, 95% CI 2-sided [64.1 to 77.9] — Treatment difference = Evolocumab QM - Placebo QM

16. Secondary Outcome: Percentage of Participants With LDL-C Less Than 70 mg/dL (1.8 mmol/L) at Week 12
Time Frame: Week 12
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 164 | 160 | 325 | 332
percentage of participants | 20.9 [15.2 to 28.2] | 21.3 [15.5 to 28.6] | 88.2 [84.0 to 91.4] | 90.2 [86.2 to 93.1]
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Cochran-Mantel Haenszel test stratified by entry statin therapy and geographic region; Treatment Difference = 67.2, 95% CI 2-sided [58.9 to 73.9] — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Cochran-Mantel Haenszel test stratified by entry statin therapy and geographic region; Treatment Difference = 68.8, 95% CI 2-sided [60.6 to 75.3] — Treatment difference = Evolocumab QM - Placebo QM

17. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) at the Mean of Weeks 10 and 12
Time Frame: Baseline and weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 164 | 160 | 325 | 332
percent change | 16.89 (17.49) | 8.48 (9.49) | -38.63 (13.67) | -42.29 (8.49)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -55.52, 95% CI 2-sided [-92.64 to -18.40], Standard Error of Mean 18.85 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -50.77, 95% CI 2-sided [-63.82 to -37.72], Standard Error of Mean 6.63 — Treatment difference = Evolocumab QM - Placebo QM

18. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) at Week 12
Time Frame: Baseline and week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 164 | 160 | 325 | 332
percent change | 26.53 (21.78) | 7.47 (10.40) | -35.93 (16.47) | -37.85 (9.02)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -62.46, 95% CI 2-sided [-110.89 to -14.03], Standard Error of Mean 24.64 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -45.32, 95% CI 2-sided [-61.87 to -28.77], Standard Error of Mean 8.42 — Treatment difference = Evolocumab QM - Placebo QM

19. Secondary Outcome: Percent Change From Baseline in Triglycerides at the Mean of Weeks 10 and 12
Time Frame: Baseline and weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 164 | 160 | 325 | 332
percent change | 11.54 (5.27) | 8.48 (4.48) | -6.48 (4.70) | -7.15 (4.02)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority; p = 0.0002, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -18.02, 95% CI 2-sided [-25.89 to -10.14], Standard Error of Mean 4.01 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -15.63, 95% CI 2-sided [-21.69 to -9.58], Standard Error of Mean 3.08 — Treatment difference = Evolocumab QM - Placebo QM

20. Secondary Outcome: Percent Change From Baseline in Triglycerides at Week 12
Time Frame: Baseline and week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 164 | 160 | 325 | 332
percent change | 10.50 (5.36) | 8.07 (4.57) | -5.91 (4.75) | -4.24 (4.09)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority; p = 0.0002, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -16.41, 95% CI 2-sided [-24.63 to -8.19], Standard Error of Mean 14.18 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -12.31, 95% CI 2-sided [-18.76 to -5.86], Standard Error of Mean 3.28 — Treatment difference = Evolocumab QM - Placebo QM

21. Secondary Outcome: Percent Change From Baseline in HDL-C at the Mean of Weeks 10 and 12
Time Frame: Baseline and weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 164 | 160 | 325 | 332
percent change | 1.25 (2.19) | 5.88 (2.11) | 7.59 (1.99) | 13.75 (1.90)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority; p = 0.0003, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 6.34, 95% CI 2-sided [3.36 to 9.33], Standard Error of Mean 1.52 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 7.87, 95% CI 2-sided [5.10 to 10.65], Standard Error of Mean 1.41 — Treatment difference = Evolocumab QM - Placebo QM

22. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 12
Time Frame: Baseline and week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 164 | 160 | 325 | 332
percent change | 2.57 (2.29) | 6.04 (2.18) | 8.45 (2.04) | 14.18 (1.95)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority; p = 0.0003, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 5.88, 95% CI 2-sided [2.49 to 9.27], Standard Error of Mean 1.72 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 8.14, 95% CI 2-sided [5.03 to 11.25], Standard Error of Mean 1.58 — Treatment difference = Evolocumab QM - Placebo QM

23. Secondary Outcome: Percent Change From Baseline in VLDL-C at the Mean of Weeks 10 and 12
Time Frame: Baseline and weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
Number analyzed (Participants) | 164 | 160 | 325 | 332
percent change | 9.63 (4.70) | 7.92 (4.43) | -17.55 (4.19) | -16.09 (3.99)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab Q2W; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -27.18, 95% CI 2-sided [-34.20 to -20.17], Standard Error of Mean 3.57 — Treatment difference = Evolocumab Q2W - Placebo Q2W
Statistical Analysis 2: Comparison: Placebo QM vs Evolocumab QM; Test type: Superiority; p < 0.0001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -24.01, 95% CI 2-sided [-29.88 to -18.14], Standard Error of Mean 2.99 — Treatment difference = Evolocumab QM - Placebo QM

ADVERSE EVENTS:
Time Frame: From the first dose of study drug to 30 days after last dose; up to 14 weeks.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Placebo Q2W | Placebo QM | Evolocumab Q2W | Evolocumab QM
All-Cause Mortality (participants affected / at risk) | 0/164 | 0/160 | 0/325 | 0/332
Serious Adverse Events (participants affected / at risk) | 6/164 | 5/160 | 10/325 | 22/332
Other Adverse Events (participants affected / at risk) | 28/164 | 22/160 | 45/325 | 49/332
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Q2W (N=164) | Placebo QM (N=160) | Evolocumab Q2W (N=325) | Evolocumab QM (N=332)
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0 | 2
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Cyst (General disorders) | 0 | 0 | 0 | 1
Herpes zoster cutaneous disseminated (Infections and infestations) | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 2 | 0
Diabetic neuropathy (Nervous system disorders) | 1 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Lacunar stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Vascular encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 1
Peripheral venous disease (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Q2W (N=164) | Placebo QM (N=160) | Evolocumab Q2W (N=325) | Evolocumab QM (N=332)
Nasopharyngitis (Infections and infestations) | 6 | 6 | 9 | 11
Upper respiratory tract infection (Infections and infestations) | 6 | 5 | 9 | 13
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 4 | 15 | 15
Hypoglycaemia (Metabolism and nutrition disorders) | 5 | 0 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1 | 6
Hypertension (Vascular disorders) | 6 | 3 | 8 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2015-11-11): https://cdn.clinicaltrials.gov/large-docs/69/NCT02662569/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/69/NCT02662569/SAP_001.pdf